CLINICAL TRIAL: NCT02093845
Title: Randomized Clinical Comparison of Everolimus-Eluting SYNERGY® and Biolimus-Eluting BioMatrix NeoFlex® Coronary Stents in Non-Selected Patients With Ischemic Heart Disease
Brief Title: Everolimus-eluting SYNERGY Stent Versus Biolimus-eluting Biomatrix NeoFlex Stent - SORT-OUT VIII
Acronym: SORT-OUT VIII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Boston Scientific Corporation (Industry); Biosensors Europe SA (Industry)
Responsible Party: Principal Investigator, Michael Mæng, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-3-14
Record Dates: First submitted 2014-02-24; First posted 2014-03-21 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
Keywords: Percutaneous coronary intervention; DES; Angina pectoris; Stent
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SYNERGY (Active Comparator): Coronary implantatation of the SYNERGY everolimus-eluting stent
  Interventions: Device: SYNERGY stent
- Biomatrix Neoflex (Active Comparator): Coronary implantation of the biolimus-eluting Biomatrix NeoFlex stent
  Interventions: Device: Biomatrix NeoFlex coronary stent

INTERVENTIONS:
Device: Biomatrix NeoFlex coronary stent — Percutaneous coronary intervention involving use of stent
  Other Names: Biolimus-eluting Biomatrix NeoFlex coronary stent
  Arms: Biomatrix Neoflex
Device: SYNERGY stent — Percutaneous coronary intervention involving use of stent
  Other Names: Everolimus-eluting SYNERGY coronary stent
  Arms: SYNERGY

SUMMARY:
The purpose of this study is to perform a randomised comparison between the SYNERGY and the Biomatrix NeoFlex stents in treatment of unselected patients with ischemic heart disease.

DETAILED DESCRIPTION:
SORT-OUT VIII is a randomised, multicenter, all-comer, two-arm, non-inferiority trial comparing the everolimus-eluting SYNERGY stent versus the Biomatrix NeoFlex stent in treatment of atherosclerotic coronary artery lesions.

Primary Endpoint:

Device-related Target Lesion Failure (TLF) hierarchically as cardiac death, non-index procedure related acute myocardial infarction (AMI) not clearly related to another lesion than the target lesion, or target lesion revascularisation (TLR) (new revascularization of target lesion) (significant stenosis in the stent ± 5 mm distal/proximal) by percutaneous coronary intervention (PCI) or coronary artery bypass operation (CABG) within 12 months.

Secondary Endpoint:

Device-related target lesion failure hierarchically as cardiac death, non-index procedure related acute myocardial infarction, not clearly related to another lesion than the target lesion, or new target lesion revascularization by percutaneous coronary intervention or coronary bypass operation at 2-5 years.

Patient-related combined endpoint hierarchically as all-cause death, non-index procedure related acute myocardial infarction or all new revascularizations by percutaneous coronary intervention or coronary bypass operation at 12, 24, 36, 48 and 60 months.

Individual above mentioned stent- or patient-related endpoints at 12, 24, 36, 48 and 60 months

MACE (combined endpoint as cardiac death, acute myocardial infarction or new revascularization of the study vessel)

Stent thrombosis defined according to the Academic Research Consortium (ARC) criteria within 24 hours (acute), between 1 and 30 days (subacute), between 30 days and 12 months (late), and after 12, 24, 36, 48 and 60 months (very late).

Device success rate defined as the frequency of a successful implantation with residual stenosis < 20% of the study stent in all the stenoses scheduled to be treated.

Procedural success rate defined as the frequency of successful implantation with residual stenosis <20% of the study stent in all the stenoses scheduled to be treated and without serious complications (cardiac death, non-index procedure related acute myocardial infarction related to target vessel or new revascularization of target lesion by percutaneous coronary intervention or coronary bypass operation).

Inclusion criteria:

All patients aged ≥18 years who are eligible for treatment with one or several drug-eluting coronary stents at one of the three heart centers in Odense, Skejby and Aalborg can be included in the study.

Exclusion criteria Age < 18 years The patient does not wish to participate The patient is not able to consent to randomization (eg intubated patients) The patient do not live in Western Denmark The patient do not speak Danish The patient is already included in this study The patient is participating in other stent studies Life expectancy <1 year Allergic to Aspirin, clopidogrel, prasugrel or ticagrelor Allergic to everolimus or biolimus Only implanted bare metal stents (BMS) Only performed plain old balloon angioplasty (POBA)

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years who are eligible for treatment with one or several drug-eluting coronary stents at one of the three heart centers in Odense, Skejby and Aalborg can be included in the study.

Exclusion Criteria:

* Age < 18 years
* The patient does not wish to participate
* The patient is not able to consent to randomization (eg intubated patients)
* The patient do not live in West Denmark
* The patient do not speak Danish
* The patient is already included in this study
* The patient is already participating in other stent studies
* Life expectancy <1 year
* Allergic to Aspirin, clopidogrel, prasugrel or ticagrelor
* Allergic to everolimus or biolimus
* Only implanted BMS
* Only performed POBA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2015-08-24 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-related target lesion failure | 12 months
  Hierarchically as cardiac death, non-index procedure related acute myocardial infarction not clearly related to another lesion than the target lesion, or target lesion revascularisation (new revascularisation of target lesion revascularisation (significant stenosis in the stent =/+ 5 mm distal/proximal) by percutaneous coronary intervention or coronary artery bypass operation

SECONDARY OUTCOMES:
Device-related target lesion failure | 2, 3, 4 and 5 years
  Hierarchically as cardiac death, non-index procedure related acute myocardial infarction not clearly related to another lesion than the target lesion, or target lesion revascularisation (new revascularisation of target lesion revascularisation by percutaneous coronary intervention or coronary artery bypass operation
Patient-related combined endpoint | 1, 2, 3, 4 and 5 year
  Hierarchically as all-cause death, non-index procedure related acute myocardial infarction, or all new revascularisation by percutaneous coronary intervention or coronary artery bypass operation
Individual above mentioned stent- or patient-related endpoints | 1, 2, 3, 4 and 5 years
MACE | 1, 2, 3, 4 and 5 years
  Combined endpoint as cardiac death, acute myocardial infarction or new revascularisation of the study vessel
Stent thrombosis | Within 24 hours, between 1 and 30 days, between 30 days and 12 months and after 1, 2, 3, 4 and 5 years
  Stent thrombosis according to the Academic Research Consortium definitions
Device success rate | intraoperative
  The frequency of a successful implantation with residual stenosis <20% of the study stent in all stenoses scheduled to be treated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maeng, MD, Principal Investigator — Aarhus University Hospital, Skejby, Aarhus N; Evald H Christiansen, MD, Study Chair — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Skejby, Aarhus N
  - Aarhus University Hospital Aalborg, Aalborg
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Maeng M, Christiansen EH, Raungaard B, Kahlert J, Terkelsen CJ, Kristensen SD, Carstensen S, Aaroe J, Jensen SE, Villadsen AB, Lassen JF, Thim T, Eftekhari A, Veien KT, Hansen KN, Junker A, Botker HE, Jensen LO; SORT OUT VIII Investigators. Everolimus-Eluting Versus Biolimus-Eluting Stents With Biodegradable Polymers in Unselected Patients Undergoing Percutaneous Coronary Intervention: A Randomized Noninferiority Trial With 1-Year Follow-Up (SORT OUT VIII Trial). JACC Cardiovasc Interv. 2019 Apr 8;12(7):624-633. doi: 10.1016/j.jcin.2018.12.036. PMID 30947936